CLINICAL TRIAL: NCT05783128
Title: The Effect of Different Methods of Airway Management on the Stomatognathic System: an Observational Prospective Study.
Status: Completed | Type: Observational
Sponsor: Aretaieio Hospital (Other)
Responsible Party: Principal Investigator, Christina Orfanou, Resident anesthesiologist, MD, MSc, Aretaieio Hospital
Other Study IDs: 453/21-09-2022
Record Dates: First submitted 2023-03-12; First posted 2023-03-24 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Airway Management; Endotracheal Intubation; Supraglottic Airway Device; Regional Anesthesia
Keywords: Intubation; Laryngeal Masks; Temporomandibular Joint Disorders; Orofacial Pain
MeSH Terms: conditions — Temporomandibular Joint Disorders; Facial Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Spontaneous breathing: 1) Spontaneous breathing, with no airway management, in surgeries performed under regional anesthesia
  Interventions: Other: Airway management techniques (exposure)
- Endotracheal intubation - Macintosh laryngoscope: 2) Assist control ventilation, after intubation through the mouth, with the use of a Macintosh laryngoscope
  Interventions: Other: Airway management techniques (exposure)
- Endotracheal intubation - C-MAC video-laryngoscope: 3) Assist control ventilation, after intubation through the mouth, with the use of a C-MAC video-laryngoscope
  Interventions: Other: Airway management techniques (exposure)
- Supraglottic Airway Device: 4) Assist control ventilation, after the insertion of an LMA (laryngeal mask airway) supreme supraglottic device
  Interventions: Other: Airway management techniques (exposure)

INTERVENTIONS:
Other: Airway management techniques (exposure) — The exposure reffers to the different methods of airway management during general or regional anesthesia.

SUMMARY:
The manipulations required during airway management and the different methods of establishing an airway (endotracheal intubation, supraglottic airway device etc) during anesthesia, as well as certain drugs used during anesthesia and sedation, may have an impact to the stomatognathic system. These effects can vary from a subtle temporomandibular joint disc displacement with reduction to the onset of temporomandibular disorders to previously healthy subjects.This observational prospective study aims at investigating the effect of different methods of airway management during anesthesia on the stomatognathic system (including temporomandibular joint, mastication muscles, occlusion etc).

DETAILED DESCRIPTION:
After being informed about the study, all patients giving written informed consent will undergo elective abdominal surgery or elective gynecological surgery (both open or laparoscopic surgeries), under general or regional anesthesia. Participants will be assigned to groups, depending on the method of airway management during anesthesia (endotracheal intubation, supraglottic airway device, sontaneous breathing).

Clinical examination of the stomatognathic system will be performed preoperatively and postoperatively (24 hours after surgery) and data concerning signs and symptoms associated with the development of temporomandibular disorders will be recorded. A follow-up questionnaire will be administered by telephone 30 days after surgery in order to record data concerning the stomatognathic system and mandibular function.

Parameters related to the physiology of the stomatognathic system, parameters related to the airway management technique, patient position, parameters related to postoperative recovery, as well as postoperative analgesic consumption will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* 18-70 years old
* ASA I-III
* elective abdominal surgery or elective gynecological surgery
* general or regional anesthesia

Exclusion Criteria:

* edentulous patients
* ear disease
* history of head and/or neck cancer
* head and neck surgery, surgery that is known to affect temporomandibular joints
* nose and/or skull base fractures
* history of dystonia/musculoskeletal disease that require treatment with muscle relaxant drugs
* cognitive impairment
* ASA > 3
* patients which underwent over 3 attempts of airway establishment during airway management
* change of anesthesia plan during surgery
* patient refusal to participate
* inability to comprehend Greek or English
* patient participation in another research project during the previous 30 days

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-70, of either sex (male, female), American Society of Anesthesiologists (ASA) physical status I-III and scheduled for elective abdominal surgery or elective gynecological surgery (both open or laparoscopic surgeries), under general or regional anesthesia, will be enrolled in the study. They will voluntarily participate in the study, have given their informed consent in writing. Participants will be assigned to groups, depending on the method of airway management during anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Pain free maximum mouth opening | 24 hours
  Assessment of maximum pain free inter-incisor distance (measured in millimeters). The examination will be conducted using the set of diagnostic tools for temporomandibular disorders (TMD), namely the Diagnostic Criteria for Temporomandibular Disorders (DC/TMD)

SECONDARY OUTCOMES:
Range of movement of the temporomandibular joint | 24 hours
  Assessement of forward and lateral movements of the jaw using the Diagnostic Criteria for Temporomandibular Disorders (DC/TMD)
Temporomandibular joint disc displacement (with/without reduction) | 24 hours
  Assessement of clicking of the jaw while opening/closing the mouth using DC/TMD
Articular sounds incidence | 24 hours
  Assessement of grinding noises and nonclassifiable sounds using DC/TMD
Subjective limitation of jaw movement | 24 hours
  Assessement of subjective report of jaw movement limitation using DC/TMD
Subjective report of orofacial pain | 24 hours
  Assessement of subjective report of orofacial pain using DC/TMD

CONTACTS AND LOCATIONS:
Overall Officials: Assosiate Professor Athanasia Tsaroucha, Study Director — Aretaieio Hospital, National and Kapodistrian University of Athens
Locations (1):
- Aretaieio Hospital, National and Kapodistrian University of Athens, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided